CLINICAL TRIAL: NCT00916630
Title: A Phase I Study of the Treatment of Recurrent Primary or Secondary CNS Lymphoma With ALIMTA (Pemetrexed), a Novel Anti-Folate
Brief Title: Treatment of Recurrent Primary or Secondary Central Nervous System (CNS) Lymphoma With ALIMTA (Pemetrexed)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Eli Lilly and Company (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jorg Dietrich, M.D., Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-097; H3-US-X059
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Central Nervous System Lymphoma
Keywords: recurrent; alimta; pemetrexed; CNS lymphoma; Primary CNS lymphoma; Metastatic lymphoma to brain
MeSH Terms: conditions — Recurrence | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm treatment (Other): Dose finding study
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — Given intravenously over a 10 to 20 minute period once every 14 days.
  Other Names: Almita

SUMMARY:
The purpose of this research study is to determine the safety of the study drug pemetrexed, and the highest dose of this drug that can be given to people safely. Another goal of this research study is to gain information about how the body handles pemetrexed and how pemetrexed may work to treat the participant's lymphoma in the nervous system. Pemetrexed (also known as Alimta) has been approved by the FDA for the treatment of some lung cancers and has been shown to be effective in laboratory studies. Information from these studies suggests that pemetrexed may help to treat patients with either primary or secondary central nervous system lymphoma.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of pemetrexed that can be given to people safely, not everyone who participates in this study will be receiving the same amount of the study drug. The dose participants will receive will depend upon the number of people that have been enrolled on the study before them and how well they have tolerated their doses of the study drug.
* Pemetrexed is given into a vein (by IV) over a 10 to 20 minute period once every 14 days. This 14 day period is called a cycle of study treatment.
* Study treatment will be divided into three phases. Induction: Participants will be given a maximum of 8 cycles. If the participant does not achieve a complete response after eight induction cycles, they will be taken off study. A complete response means there is no evidence of disease on MRI or CT scan. Consolidation: If the participant has achieved complete response, they will have two additional cycles. Maintenance: Following the completion of the consolidation cycles, participants will receive the study drug only once per month. They can continue to receive maintenance cycles for up to a year from the start of the first induction cycle.
* Folic acid and vitamin B12 are two vitamins that have been shown to help lessen the severity of some side effects of pemetrexed. Participants will begin taking oral folic acid tablets at least 5 days before their first dose of pemetrexed and daily until 3 weeks after their last dose. Vitamin B12 is given through injections into your muscle. Participants will receive their first vitamin B12 injection 1-2 weeks before their first dose of pemetrexed. They will receive injections every 9 weeks.
* Corticosteroids such as dexamethasone have been shown to help prevent severe skin rashes associated with pemetrexed. Participants will receive dexamethasone twice daily starting the day before each pemetrexed infusion continuing until the day after each infusion.
* On day 1 of each cycle the following will be performed: a physical examination, blood work, vital signs, assessment of who well the participant is functioning, and mini-mental examination. On day 8 of each cycle blood work will be performed.
* Research blood work will be obtained (PKs) over the first four days of cycles 1 and 2 (or study participation days 1-4 and 15-18).
* Participants will come to the clinic once a month during the maintenance cycles for a physical examination, blood work, assessment of how well the participant is functioning, vital signs and mini-mental examination.
* Tumor assessments by MRI will be done after every 2 cycles during the induction and consolidation cycles. During the maintenance cycles the MRIs will be repeated every 2 cycles (once every 2 months).
* Collection of cerebral spinal fluid (CSF) for research tests will also likely be performed, if safe for you, to learn more about how well pemetrexed can cross the blood-brain barrier. This will be performed by one of two methods 6 and 24 hours after the pemetrexed is infused on days 1 and 2 of the first two cycles.
* After Alimta is given you will also receive, a white blood cell recruiting material, Neupogen to avoid suppressing your bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Disease state (5 categories of patients with these extremely rare disease are eligible: 1) Patients intolerant of Methotrexate-must have a diagnosis of B cell non-Hodgkin's lymphoma 2) Patients unable to receive methotrexate due to lack of drug availability-must have a diagnosis of B cell non-Hodgkin's lymphoma 3) Patients who fail to achieve a complete response to initial therapy for primary CNS lymphoma-must have a diagnosis of B cell non-Hodgkin's lymphoma 4) Recurrent Primary CNS lymphoma-If in the judgement of the treating physician therapy would be initiated without a repeat biopsy then the original biopsy with a diagnosis of B cell non-Hodgkin's lymphoma will suffice 5) Secondary CNS lymphoma-If in the judgement of the treating physician therapy would be initiated without a repeat biopsy then the original biopsy with a histologic diagnosis of B cell non-Hodgkin's lymphoma will suffice.
* Histologic diagnosis of B cell non-Hodgkin's lymphoma with measurable disease OR cytologic diagnosis of B cell non-Hodgkin's lymphoma with measurable disease OR immunohistochemical diagnosis of monoclonality (CDF) with or without measurable intracranial disease OR molecular diagnostic diagnosis of monoclonality CSF) with or without measurable intracranial disease OR Ocular-patients may have a combination of histologic confirmation of ocular lymphoma and measurable intracranial tumor. Slit-lamp examination and vitreal or retinal biopsy will be done to confirm ocular lymphoma OR neurolymphomatosis-evidence of measurable disease as nerve seeking lymphoma on MRI imaging with histologic diagnosis at any site.
* Karnofsky score of 60 or greater
* Must be able to undergo MRI scanning
* 18 years of age or older
* Life expectancy of at least 2 months
* Laboratory values as outlined in protocol
* Must be willing to practice an effective method of birth control during participation in the study whether male or female.

Exclusion Criteria:

* Definitive histologic diagnosis of low grade lymphoma without substantive clinical suspicion of transformation to an aggressive lymphoma
* Renal dysfunction defined as creatinine clearance < 45 ml/min or serum creatinine > 2mg/dL
* Transaminases > 3 times above the upper limits of the institutional normal
* Acute infection, granulocytopenia or medical condition precluding surgery as judged by the caring physician and review team
* Pregnant or lactating females
* Patients must not have pre-existing immunosuppression, concurrent immunosuppressive treatment (with the exception of dexamethasone) or be a transplant recipient
* Patients must not have received prior whole brain irradiation. They can have received prior focal irradiation
* Prior participation in chemotherapy, cytotoxic therapy, immunotherapy or therapeutic protocols within 4 weeks fo enrollment. Patients unable to stop NSAIDS or Cox 2 inhibitors for two day before and after treatment as well as the day of treatment
* No other active systemic malignancy with the exception of basal cell carcinoma of the skin and cervical carcinoma in situ. Patients with a remote history (5 years or more) of malignancy are eligible for the protocol in the absence of active disease
* Clinically relevant third space fluid collection refractory to drainage
* Patient refusal to participate in the pK study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and to determine the maximum tolerated dose of pemetrexed given intravenously for the treatment of recurrent lymphoma invading the CNS. | 6 years

SECONDARY OUTCOMES:
To determine the plasma pharmacokinetics of pemetrexed and assess drug penetration into the CSF. | 6 and 1/2 years
To provide preliminary evidence of pemetrexed activity against brain lymphoma my MRI criteria of clearance of CSF lymphoma cells. | 6 years
To identify the time to complete response. | 6 years
To provide a measure of reduction of enhancing tumor volume as compared to our nomogram of reduction of tumor volume for methotrexate recipients with brain lymphoma. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Dietrich, MD PhD MMSc, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts